CLINICAL TRIAL: NCT06849232
Title: A COMPARATIVE STUDY of PLATELET-RICH PLASMA and NORMAL SALINE DRESSINGS in the TREATMENT of CHRONIC WOUNDS
Brief Title: A Comparative Study of Platelet-Rich Plasma and Normal Saline Dressings in the Treatment of Chronic Wounds (PRP-NS Wound T)
Acronym: PRP-NS Wound T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quaid-e-Azam Medical College (Other)
Responsible Party: Principal Investigator, Shahid Hussain, Associate Professor of Surgery, Quaid-e-Azam Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2381/DME/QAMC Bahawalpur; 2381/DME/QAMC (Other: Department of medical education, QAMC Bahawalpur)
Record Dates: First submitted 2025-02-08; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Wound Healing
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRP Dressing Group (Experimental): wounds were first cleaned with normal saline, followed by the injection of PRP, prepared from the patient's own blood by the hematology department, into the surrounding wound area twice weekly
  Interventions: Procedure: Platelet-Rich Plasma (PRP) Injections
- Normal Saline Dressing Group (Active Comparator)
  Interventions: Procedure: Platelet-Rich Plasma (PRP) Injections

INTERVENTIONS:
Procedure: Platelet-Rich Plasma (PRP) Injections — wounds were first cleaned with normal saline, followed by the injection of PRP, prepared from the patient's own blood by the hematology department, into the surrounding wound area twice weekly

SUMMARY:
This study aims to compare the effectiveness of Platelet-Rich Plasma (PRP) dressings versus Normal Saline dressings in the treatment of chronic wounds. Chronic wounds are slow-healing wounds that can cause significant discomfort, increase the risk of infections, and impact a patient's quality of life.

Platelet-Rich Plasma (PRP) is derived from the patient's own blood and contains growth factors that may help promote faster wound healing. On the other hand, Normal Saline dressings are commonly used as a standard wound care approach.

Participants in this study will be randomly assigned to receive either PRP dressings or normal saline dressings. The healing progress of their wounds will be monitored over a specified period to determine which treatment leads to better and faster healing.

The findings from this study may help improve wound care management and provide evidence for using PRP as an effective treatment for chronic wounds.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-60 years of either gender were included if they had a chronic wound persisting for at least six weeks and with a size of at least 2 × 2 cm.

Exclusion Criteria:

* Patients were excluded if their wounds had existed for less than six weeks, if they had a previous history of PRP dressing use, or if they had documented hypersensitivity to PRP.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 156 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
Wound Healing Rate | April 17, 2024, to October 16, 2024

CONTACTS AND LOCATIONS:
Locations (1):
- Bahawal Victoria Hospital, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No